CLINICAL TRIAL: NCT04921397
Title: China Stroke Registry for Patients With Traditional Chinese Medicine (CASES-TCM): A Prospective, Multicenter, Observational Study
Brief Title: China Stroke Registry for Patients With Traditional Chinese Medicine
Acronym: CASES-TCM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Ying Gao, President of Institute for Brain Disorders, Beijing University of Chinese Medicine, Dongzhimen Hospital, Beijing
Other Study IDs: 2021XS-001
Record Dates: First submitted 2021-06-01; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Ischemic Stroke; Intracerebral Hemorrhage
MeSH Terms: conditions — Ischemic Stroke; Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The CASES-TCM study is a prospective, multicenter, observational study, which will enroll 20,000 patients with acute stroke (ischemic stroke or intracerebral hemorrhage) within 7 days of symptom onset.

This study attempts to depict major clinical characteristics of acute stroke in patients with Chinese medicine treatment and to explore any difference compared with other non-Chinese medicine use cohorts and the effectiveness and safety of Chinese medicine.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Diagnosed as acute ischemic stroke or intracerebral hemorrhage
* Within 7 days of symptom onset

Exclusion Criteria:

* Refusal to give informed consent
* Have difficulties completing follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet the criteria will be consecutively enrolled from 100 participating sites in China.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2021-06-11 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Distribution of scores on the modified Rankin scale at 3-month follow-up | 3 months follow-up
  Modified Rankin Scale, a commonly used scale for measuring the degree of dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. 0 - No symptoms.1 -No significant disability. Able to carry out all usual activities, despite some symptoms.2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.3 - Moderate disability. Requires some help, but able to walk unassisted.4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.6 - Dead.
Recurrent stroke events (ischemic stroke, hemorrhagic stroke including intracerebral hemorrhage and subarachnoid hemorrhage) within 12-month follow-up | 12 months follow-up
  Number of patients with new ischemic stroke and hemorrhagic stroke within 12 months of follow-up.

SECONDARY OUTCOMES:
Proportion of patients receive Chinese medicine treatment within 24 hours after admission | 24 hours after admission
  Chinese medicine treatment exposure defined as whether patients receive Chinese medicine injection, oral Chinese patent medicine, or compound Chinese medicine.
Chinese medicine treatment duration within 3-month, 12-month, and 24-month follow-up | 3 months, 12 months, and 24 months follow-up
  Chinese medicine treatment duration will be assessed using proportion of days covered, which is a percentage of days covered with the medicine in the number of days the patient is eligible to have the medication.
Change in the National Institutes of Health Stroke Scale score between baseline (admission) and discharge | At admission (baseline) and discharge (14 days - mean for length of hospitalization for stroke patients)
  National Institute of Health Stroke Scale is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. It is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
Patient-Reported Outcomes Scale for Stroke score at discharge | At discharge (14 days - mean for length of hospitalization for stroke patients)
  Patient-Reported Outcomes Scale for Stroke, a structured questionnaire-scale was developed suitable for Chinese patients. The score ranges from 0 (best) to 144 (worst).
Proportion of patients with modified Rankin Scale score ≤2 at 3-month and 12-month follow-up | 3 months, 12 months follow-up
  Modified Rankin Scale, a commonly used scale for measuring the degree of dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. 0 - No symptoms.1 -No significant disability. Able to carry out all usual activities, despite some symptoms.2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.3 - Moderate disability. Requires some help, but able to walk unassisted.4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.6 - Dead.
Distribution of scores on the modified Rankin scale at 12-month follow-up | 12 months follow-up
  Modified Rankin Scale, a commonly used scale for measuring the degree of dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. 0 - No symptoms.1 -No significant disability. Able to carry out all usual activities, despite some symptoms.2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.3 - Moderate disability. Requires some help, but able to walk unassisted.4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.6 - Dead.
Proportion of patients with Barthel Index score ≥90 at 3-month and 12-month follow-up | 3 months, 12 months follow-up
  Barthel Index is a commonly used scale for measuring the activity of daily living of people. Score of 10-item scale ranges from 0 (worst) to 100 (best).
Recurrent stroke events (ischemic stroke, hemorrhagic stroke including intracerebral hemorrhage and subarachnoid hemorrhage) within 3-month and 24-month follow-up | 3 months, 24 months follow-up
  Number of patients with new ischemic stroke and hemorrhagic stroke events within 3 months and 24 months of follow-up.
Composite of new clinical vascular events within 3-month, 12-month, and 24-month follow-up | 3 months, 12 months, 24 months follow-up
  Number of patients with new clinical vascular events (ischemic stroke/ hemorrhagic stroke/ transient ischemic attack / myocardial infarction /vascular death) within 3 months, 12 months, and 24 months of follow-up.
Mini-Mental State Examination scale score at 3-month, 12-month, and 24-month follow-up | 3 months, 12 months, 24 months follow-up
  Mini-Mental State Examination scale is a commonly used scale for measuring the cognitive function. Range: 0 to 30 points, higher points represent a better outcome.
All-cause mortality within 12-month and 24-month follow-up | 12 months, 24 months follow-up
  Number of patients who died within 12 months and 24 months of follow-up.
Incidence of adverse events | Up to 24 months follow-up
  Number of patients with any adverse events (including serious adverse events) during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Gao, Principal Investigator — Dongzhimen Hospital, Beijing
Locations (1):
- Dongzhimen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feng L, Kong L, Dong X, Lai X, Zhang D, Ren B, Liu S, Xie X, Li C, Song Y, Du Y, Cao K, Zhang C, Gao Y; CASES-TCM Protocol Steering Group. China Stroke Registry for Patients With Traditional Chinese Medicine (CASES-TCM): Rationale and Design of a Prospective, Multicenter, Observational Study. Front Pharmacol. 2021 Aug 31;12:743883. doi: 10.3389/fphar.2021.743883. eCollection 2021. PMID 34531755